## **Final Statistical Analysis Plan for:**

#### NCT03009058

Study IMM-101-011

A Novel Phase I/IIa Open-label Study of IMM-101 in Combination with Selected Standard of Care (SOC) Regimens in Patients with Metastatic Cancer or Unresectable Cancer at Study Entry

# Statistical Analysis Plan

## **Immodulon Therapeutics Limited**

Protocol: IMM-101-011

**Treatment: IMM-101** 

A Novel Phase I/IIa Open-label Study of IMM-101 in Combination with Selected Standard of Care Regimens in Patients with Metastatic Cancer or Unresectable Cancer at Study Entry

Author: Statistical

Consultant on behalf of Immodulon Therapeutics Limited

Document Status: Final V1.0

Version Date: 26 September 2017

#### STATEMENT OF CONFIDENTIALITY

This document contains information confidential and/or of proprietary interest to Immodulon Therapeutics Limited. No part of this document may be copied or disclosed to a third party in any format (including oral, printed, written or electronic), without the written permission of Immodulon Therapeutics Limited, except insofar as it is necessary for assessment by appropriate bodies such as ethics committees or regulatory authorities under the same conditions of confidentiality. It must be returned to Immodulon Therapeutics Limited upon request.

# **Approvals**

Author:



26Sep2017 **Date** 

on benan of immodulon Therapeutics Ltd

Reviewer:



26 SEP 2017 Date

Approved by:



26 - Scp - 2017 Date

# **Contents**

| 2 Abbreviations | 4 |
|-----------------------------------------------------------------------|----|
| 3 Introduction | 5 |
| 3.1 Protocol Status and Termination by Immodulon | |
| 4 Study Objectives | 6 |
| 5 Study Design | 6 |
| 5.1 Study Schedule | 6 |
| 5.1.1 Flowchart of Assessments: Screening and Treatment Phases | 7 |
| 5.1.3 Flowchart of Assessments: Long-term Maintenance Treatment Phase | 11 |
| 5.2 Study Data Sets | 13 |
| 5.2.1 All Enrolled Patients | 13 |
| 5.2.2 Safety Analysis Set (SAF) | 13 |
| 5.3 Withdrawn Patients | 13 |
| 5.4 Randomisation | 13 |
| 5.5 Blinding | 13 |
| 5.6 Sample Size | 13 |
| 5.7 Changes in Conduct or Planned Analyses from the Protocol | 13 |
| 6 Statistical Methodology | 13 |
| 6.1 Planned Presentations of Data: Listings | |
| 6.1.1 Standard Calculations | 14 |
| 6.2 Adjustment for Covariates | 20 |
| 6.2.1 Centre Effects | 20 |
| 6.3 Protocol Violations | |
| 6.4 Missing Values – Missing Visits | 20 |
| 6.5 Deviations from Statistical Analysis Plan | 20 |

## 2 Abbreviations

| AE | Adverse Event |
|-----------|------------------------------------------------------------------|
| ATC | Anatomical Therapeutic Chemical |
| eCRF | Electronic Case Report Form |
| CSR | Clinical Study Report |
| Immodulon | Immodulon Therapeutics Limited |
| irRC | Immune-related response criteria |
| 011 study | IMM-101-011 study |
| MedDRA | Medical Dictionary for Regulatory Activities |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SAF | Safety Analysis Set (All randomised patients from the Main Study |
| | who receive at least one dose of study drug) |
| SQN | Syne qua non Ltd |
| SOC | Standard of Care |
| WHO | World Health Organisation |

#### 3 Introduction

This document presents the statistical analysis plan (SAP) for Immodulon Therapeutics Limited (Immodulon), Protocol No. IMM-101-011: A Novel Phase I/IIa Open-label Study of IMM-101 in Combination with Selected Standard of Care Regimens in Patients with Metastatic Cancer or Unresectable Cancer at Study Entry.

### 3.1 Protocol Status and Termination by Immodulon

On 31<sup>st</sup> July 2017, Immodulon took the decision to enroll no further patients into this Phase I/IIa open-label study and to close the study early.

On 31<sup>st</sup> July 2017, 2 patients were on study and 1 patient was a screen failure. Both enrolled patients were consented into Cohort 6 (IMM-101 + Anti-PDI (Pembrolizumab, Nivolumab) in metastatic melanoma). For these 2 treated patients the last study visit completed was Visit 5 – Week 10. The End of Study / Withdrawal Visit was completed in place of Visit 6 – Week 12 for both patients.

It was planned to evaluate up to 20 patients in each SOC (standard of care)/tumour type, with a total of approximately 300 patients enrolled overall (across 7 tumour types), with assessment of both safety and efficacy by each SOC/tumour type. Further details of the sample size evaluations are given in the study protocol. A minimum of 10 patients per cohort were required for an evaluation of futility with respect to the primary activity endpoint of response to treatment (based on immune-related response criteria [irRC]). Given that only two patients were enrolled into the study, the objectives of the study described in the study protocol cannot be met.

The planned statistical analysis described in the study Protocol will not now be performed due to the early closure of the study. However all clinical study data will be presented in data listings, as described in this statistical analysis plan (SAP) and in the separate document containing detailed Planned Listings Shells. Both documents will be approved before database lock. The listings will be produced in accordance with the approved Listings Shells, by Syne qua non Ltd (SQN) (SQN Study No: ICS16001).

This analysis plan is based on the final protocol version 4 (released 25 October 2016) and the final 011 study electronic case report form (eCRF), version 4, dated 3 March 2017. Given the early termination of the study, this SAP is therefore abbreviated. Relevant sections of the study Protocol are referred to and for ease of reference, the full study activity schedule is reproduced from the study Protocol.

### 4 Study Objectives

Full details of the study objectives, endpoints and evaluation methodology are given in the study Protocol.

#### 5 Study Design

Full details of the study design are provided in the study Protocol.

### 5.1 Study Schedule

For the 2 patients enrolled into the study, the last study visit completed was Visit 5 – Week 10. The End of Study / Withdrawal Visit was completed in place of Visit 6 – Week 12 for both patients.

The study schedule of assessments is presented in Sections 5.1.1 and 5.1.2. Note that a number of inconsistencies within the study Protocol version 4.0 were noted by Immodulon (file note IMM/011/FN/0008), approved 16 Mar 2017, as follows:-

- The screening phase was between Day -28 to Day -1 (not Day -7 as indicated in the Protocol version 4.0 study schedule of assessments)
- The response to treatment was to be assessed at Weeks 6 and 10 and End of Study/Withdrawal Visit (this was omitted from the assessment schedule in error)
- Footnote 42 (Screening and Treatment phases) and 21 (Long-term maintenance phase): Full text was amended to 'Solicited and visible injection site reactions will be recorded and patients will be asked to assess any impact on their daily activities and whether the reactions are getting better, worse or staying the same. (The question asked was omitted from the assessment schedule in error).

# **5.1.1 Flowchart of Assessments: Screening and Treatment Phases**

| | Screening<br>Phase | | Treatment Phase | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Week -4/-1 | Week 0 | Week 2 | Week 4 | Week 8 | Week 10 | Week 12 | Week 16 | Week 20 | Week 24 | Week 28 |
| Day | Day -28 to -7 | Day 0 | Day 14 | Day 28 | Day 56 | <b>Day 70</b> | Day 84 | <b>Day 112</b> | Day 140 | Day 168 | Day 196 |
| , | | Visit 1 | Visit 2 | Visit 3 | Visit 4 | Visit 5 | Visit 6 | Visit 7 | Visit 8 | Visit 9 | Visit 10 |
| Visit window (days) | - | - | | | ±3 days[1] | | | | ±14 d | ays[1] | |
| Informed consent[2] | ✓ | | | | | | | | | | |
| Inclusion/exclusion criteria | ✓ | <b>√</b> [3] | | | | | | | | | |
| Demography & baseline data[4] | ✓ | | | | | | | | | | |
| Complete medical history[5] | ✓ | | | | | | | | | | |
| Physical examination[6] | ✓ | | | | | | | | | | ✓ |
| Safety blood and serum samples[7,8] | <b>√</b> [9,10,11] | <b>√</b> [11] | <b>√</b> [11,12] | <b>√</b> [11,12] | <b>√</b> [11,12] | <b>√</b> [11,12] | <b>√</b> [11,12] | <b>√</b> [11] | <b>√</b> [11] | <b>√</b> [11] | <b>√</b> [11,12] |
| HLA serotyping[13] | ✓ | | | | | | | | | | |
| Immunomarkers[14] | <b>√</b> [9] | | | | | | <b>√</b> [12] | | | <b>√</b> [12] | |
| Serum pregnancy test[15] | ✓ | | | | | | | | | | |
| Vital signs[16] | ✓ | <b>√</b> [17] | | | | | | | | | ✓ |
| Weight | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ |
| 12-lead ECG[18] | ✓ | | | | | | | | | | |
| ECOG/WHO performance status[19] | <b>√</b> [20] | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ |
| Tumour biopsy - slides[21,22] | <b>√</b> [23] | | | | | | | | | | <b>√</b> [24,25] |
| Tumour biopsy – core samples [22,26] | <b>√</b> [27,28] | | | | <b>√</b> [25,29] | | | | | | <b>√</b> [25,29] |
| Microsatellite phenotyping[30] | ✓ | | | | | | | | | | |
| CT/MRI scan | <b>√</b> [31] | | | | | | <b>√</b> [32] | | | | <b>√</b> [32] |
| Measure diameter of erythema and skin biopsy[26,27,33,34] | | | <b>√</b> [35,36] | | <b>√</b> [35,36] | | | | | | <b>√</b> [35,36] |

Final Version 1.0  26Sept2017

| | Screening<br>Phase | | Treatment Phase | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Week -4/-1 | Week 0 | Week 2 | Week 4 | Week 8 | Week 10 | Week 12 | Week 16 | Week 20 | Week 24 | Week 28 |
| Day | Day -28 to -7 | Day 0 | Day 14 | <b>Day 28</b> | Day 56 | Day 70 | Day 84 | Day 112 | Day 140 | Day 168 | Day 196 |
| Day | Day -26 to -7 | Visit 1 | Visit 2 | Visit 3 | Visit 4 | Visit 5 | Visit 6 | Visit 7 | Visit 8 | Visit 9 | Visit 10 |
| Visit window (days) | - | - | ±3 days <sup>[1]</sup> | | | | ±14 days <sup>[1]</sup> | | | | |
| Prior/concomitant therapy[37] | <b>√</b> [38] | <b>√</b> [38] | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ |
| Adverse event reporting[39] | <b>√</b> [40] | <b>√</b> [41] | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ |
| Assess injection site reactions[12] | | | √[42] | <b>√</b> [42] | <b>√</b> [42] | <b>√</b> [42] | <b>√</b> [42] | <b>√</b> [42] | <b>√</b> [42] | <b>√</b> [42] | <b>√</b> [42] |
| Record time interval since last dose of IMM-101[1,12] | | | <b>√</b> | ✓ | ✓ | ✓ | <b>√</b> | <b>✓</b> | <b>✓</b> | ✓ | ✓ |
| Check time interval since last dose of IMM-101 is $\ge$ 11 days (14 days $\pm$ 3 days)[1,12] | | | <b>√</b> | ✓ | <b>√</b> | <b>√</b> | <b>√</b> | | | | |
| IMM-101 administration | | <b>√</b> [41] | <b>√</b> [43] | ✓ | ✓ | <b>√</b> [43] | ✓ | ✓ | ✓ | ✓ | ✓ |

#### **Footnotes:**

ALP: alkaline phosphatase; ALT: alanine transaminase; AST: aspartate transaminase; β-hCG: β-human chorionic gonadotropin; BCG: Bacillus Calmette–Guérin; CA19.9: carbohydrate antigen 19.9; CEA: carcinoembryonic antigen; CKD-EPI: Chronic Kidney Disease Epidemiology Collaboration; CRP: C-reactive protein; CT: computerised tomography; ECG: Electrocardiogram; ECOG: Eastern Cooperative Oncology Group; eCRF: electronic case report form; eGFR: estimated glomerular filtration rate; FACS: fluorescence-activated cell sorting; FBC: full blood count; GEM: gemcitabine; GGT: gamma-glutamyl transferase; Hb: haemoglobin; HLA: human leukocyte antigen; INR: international normalised ratio; LDH: lactate dehydrogenase; LFT: liver function test; MCH: mean cell haemoglobin; MCV: mean cell volume; miRNA: micro ribonucleic acid; MPV: Mean platelet volume; MRI: magnetic resonance imaging; Pt: prothrombin time; PTT: partial thromboplastin time; RBC: red blood cell; WBC: white blood cell; WHO: World Health Organisation.

- 1. During the Treatment Phase of the study (Doses 1 to 3 and Doses 4 to 6), at the discretion of the Investigator, the dose interval may be modified provided the minimum period between doses is at least 11 days (14±3 days). However, in the event that this minimum dosing interval cannot be maintained, at the discretion of the Investigator, a half dose of IMM-101 (0.5 mg/0.05 mL intradermal injection) should be given and at no point in the study should any doses of IMM-101 be administered at less than a 7-day interval. Where this reduced dosing interval is being used the 4-week interval between Dose 3 and Dose 4 and between Dose 6 and Dose 7 should still be maintained. In the event of an injection site reaction of ≥Grade 3 (severe) as measured by the NCI CTCAE v4.0, at the discretion of the Investigator, patients may be administered a half dose of IMM-101 (i.e., a single 0.05 mL intradermal injection of IMM-101).
- 2. Before beginning any study procedure, the patient will read and sign an informed consent form. The patient will be given a copy of the signed informed consent form.


- 3. Inclusion/exclusion criteria will be re-checked before commencing any study treatment including confirmation of anticipated life expectancy ≥3 months and a review of blood and serum samples. Final determination of patient eligibility will be made upon receipt of all clinical laboratory results and assessment of all inclusion and exclusion criteria.
- 4. Gender, date of birth, ethnicity and height.
- 5. Full medical history including disease history and treatment, any concurrent illnesses and history of previous injections (e.g. smallpox, yellow fever, BCG).
- 6. A full physical examination will be performed, including assessment of injections received prior to Screening and pre-existing injection site reactions (i.e. BCG or prior cancer treatment reactions). Any additional physical examinations to those scheduled for this study will be performed as per the Investigator's routine procedures.
- 7. Blood and serum samples (6 mL blood) CRP, FBC (Hb, Haematocrit, RBC count, WBC count, WBC differential count, platelet count, MPV, MCV, MCH), LFTs (ALT, ALP, AST, bilirubin [total, direct], albumin, total protein, GGT, Pt/PTT, INR, LDH), calcium, urea and electrolytes (kidney function: sodium, potassium, creatinine, urea, eGFR [using CKD-EPI creatinine calculation]), CEA, CA19.9.
- 8. Any additional blood tests to those scheduled will be performed as per the Investigator's routine procedures.
- 9. Screening blood tests should be taken within 7 days prior to the start of the study.
- 10. Review of blood test results: Screening blood test results must be available at least 24 hours prior to IMM-101 administration.
- 11. Patients in the anti-PD1 and anti-CTLA-4 cohorts only, prior to every course of checkpoint inhibitor as per the label: thyroid function test; ACTH; blood glucose test; lipase.
- 12. Prior to administration of IMM-101.
- 13. 4 mL whole blood (Only needs to be taken if the result is not already available for the patient).
- 14. Immunological markers:
  - 6 mL whole blood: miRNA panel, circulating metabolites.
  - 6 mL whole blood will be collected from a subset of patients for FACS analysis: immune cell quantification.
  - 6 mL whole blood will be collected from a subset of patients to be analysed in the TruCulture system: cytokines, chemokines, immune mediators; functional immune cell assays, tumour markers.
- 15. A Screening serum pregnancy test (β-hCG) will be performed on all eligible female patients of child bearing potential within 72 hours prior to the start of the study. A negative serum pregnancy test result must be obtained prior to a female patient of child bearing potential receiving study medication. Serum pregnancy tests should be repeated as warranted during the study.
- 16. Resting blood pressure, pulse, and body temperature will be recorded as vital signs. Additional measures of vital signs to those scheduled for this study will be performed as per the Investigator's routine procedures.
- 17. Patients should be followed by vital sign monitoring for at least 2 hours after administration of IMM-101, under medical supervision with resuscitation facilities available as a precautionary measure.
- 18. 12-lead ECG measures will be recorded at Screening. Additional 12-lead ECG measures to those scheduled for this study will be performed as per the Investigator's routine procedures.
- 19. Two observers will be required to assess performance status. If there is any discrepancy between the two scores, the highest (worst) assessment will be used
- 20. To be eligible for inclusion in the study, patients must have an ECOG/WHO performance status of  $\leq 2$  at Day 0.
- 21. Not for patients with metastatic pancreatic cancer who will receive GEM monotherapy, and patients with metastatic melanoma who will receive a PD1 checkpoint inhibitor
- 22. Any trauma and clinical sequelae related to the mechanics of the tumour biopsy should be reported as related to the study procedure
- 23. Document results and record the date of the last tumour biopsy on the patient's eCRF.


- -For patients receiving first line treatment, if no biopsy has been performed in the 3 months prior to Screening, a biopsy should be performed during the Screening period, or at Day 0, when eligibility has been confirmed and before first dose of IMM-101 is administered and 10 anonymised, unstained slides prepared from the diagnostic specimen (any additional biopsies to those scheduled for this study will be performed as per the Investigator's routine procedures).
- -For patients receiving second, third and fourth line treatment, if no biopsy has been performed in the 2 years prior to Screening a biopsy should be performed during the Screening period, or at Day 0, when eligibility has been confirmed and before first dose of IMM-101 is administered and 10 anonymised, unstained slides prepared (any additional biopsies to those scheduled for this study will be performed as per the Investigator's routine procedures).
- 24. This tumour biopsy is optional and undertaken only if the patient provides consent for it.
- 25. The Investigator will schedule the biopsy at this visit. The biopsy will be performed within 2 weeks after this visit
- 26. Only in patients with metastatic pancreatic cancer who will receive GEM monotherapy, and patients with metastatic melanoma who will receive a PD1 checkpoint inhibitor
- 27. The Investigator will select the lesion to be biopsied, on the basis of a lesion that will be the most feasible to access and which provides the lowest risk to the patient. Three core biopsy samples will be taken from the target lesion and prepared as follows: 1 core snap frozen, 1 core paraffin embedded, 1 core cryoblock.
- 28. These patients will undergo a tumour biopsy during the Screening period, or at Day 0, when eligibility has been confirmed and before first dose of IMM-101 is administered.
- 29. The Investigator will biopsy the same lesion that was biopsied at Screening
- 30. For patients with colorectal cancer only (if not already available for the patient)
- 31. Document results and record date of last CT/MRI scan on the patient's eCRF. If no scan has been performed in the 30 days prior to Screening a scan should be performed.
- 32. Scans performed to assess progression or response must match the baseline scan (i.e. if CT scan at baseline then CT scan for all other scans). Additional CT/MRI scans to those scheduled for this study will be performed as per the Investigator's routine procedures.
- 33. Prior to administration of IMM-101
- 34. Length and width
- 35. From the arm into which the previous dose was administered
- 36. Skin punch biopsy reactions assessed at the following visit. Any trauma and clinical sequelae related to the mechanics of the skin biopsy should be reported as related to the study procedure and not reported as an injection site reaction.
- 37. All prescription and over-the-counter medications, including herbals, homeopathic remedies etc., will be recorded.
- 38. Record any prior/concomitant therapy/medications taken up to 4 weeks before initiation of Screening and any prior/concomitant depot corticosteroids taken up to 6 weeks before initiation of Screening
- 39. All AEs will be followed until resolution, death, or 30 days after the Withdrawal/EOS visit (whichever comes first)
- 40. Pre-existing conditions will be recorded.
- 41. Patients will be observed for 2 hours post dose, prior to leaving the study site.
- 42. Solicited and visible injection site reactions will be recorded.
- 43. Patients receiving the reduced intensity IMM-101 dosing regimen will not receive IMM-101 at this visit.


## 5.1.3 Flowchart of Assessments: Long-term Maintenance Treatment Phase

| | | | | | | | | | | End of | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Nominal Time Point | Week 32 | Week 36 | Week 40 | Week 44 | Week 48 | Week 52[1] | Week 56 | Week 60 | Week 64 | Week 68 | Week<br>nn[2,3] | Study/<br>With-<br>drawal |
| Visit/Dose | Visit 11 | Visit 12 | Visit 13 | Visit 14 | Visit 15 | Visit 16 | Visit 17 | Visit 18 | Visit 19 | Visit 20 | Visit nn | Visit[4] |
| Visit window (days) | | | | | | ±14 d | ays[5] | | | | | |
| Physical examination[6] | | | | | | | | | | | | ✓ |
| Safety blood and serum samples[7,8,9] | <b>√</b> [10] | <b>√</b> [10,11] | <b>√</b> [10] | <b>√</b> [10] | <b>✓</b> [10,11] | <b>√</b> [10] | <b>√</b> [10] | <b>√</b> [10,11] | <b>√</b> [10] | <b>√</b> [10] | <b>√</b> [10,11] | <b>√</b> [12] |
| Immunomarkers[8,13] | | <b>√</b> [11] | | | <b>√</b> [11] | | | <b>√</b> [11] | | | <b>√</b> [11] | ✓ |
| Vital signs[14] | | | | | | | | | | | | <b>√</b> [14] |
| Weight | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ |
| 12-lead ECG[15] | | | | | | | | | | | | ✓ |
| ECOG/WHO performance status[16] | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ |
| CT/MRI scan[17] | | | | | | | | | | | | <b>√</b> [18] |
| Prior/concomitant therapy[19] | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ |
| Adverse event reporting[20] | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ |
| Assess injection site reactions[8,21] | <b>✓</b> | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | <b>✓</b> | ✓ |
| Record time interval since last dose of IMM-101[5,8] | ✓ | <b>✓</b> | <b>✓</b> | ✓ | <b>~</b> | ✓ | ✓ | <b>~</b> | <b>✓</b> | <b>✓</b> | <b>~</b> | |
| IMM-101 administration | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | |

#### **Footnotes:**

ALP: alkaline phosphatase; ALT: alanine transaminase; AST: aspartate transaminase; CA19.9: carbohydrate antigen 19.9; CEA: carcinoembryonic antigen; CKD-EPI: Chronic Kidney Disease Epidemiology Collaboration; CRP: C-reactive protein; CT: computerised tomography; ECG: Electrocardiogram; ECOG: Eastern Cooperative Oncology Group; eGFR: estimated glomerular filtration rate; EOS: End of Study; FACS: fluorescence-activated cell sorting; FBC: full blood count; GGT: gamma-glutamyl transferase; Hb: haemoglobin; INR: international normalised ratio; LDH: lactate dehydrogenase; LFT: liver function test; MCH: mean cell haemoglobin; MCV: mean cell volume; miRNA: micro ribonucleic acid; MPV: Mean platelet volume; MRI: magnetic resonance imaging; Pt: prothrombin time; PTT: partial thromboplastin time; RBC: red blood cell; WBC: white blood cell; WHO: World Health Organisation.


- 1. A reduction in dose and/or an increase in the dosing interval may be required after one year
- 2. Should the study extend beyond 68 weeks, the same pattern of assessments will continue for subsequent visits as described in this Schedule of Assessments.
- 3. A reduction in dose and/or an increase in the dosing interval may be required after one year.
- 4. Patients withdrawing from the study at any time should attend this EOS visit within 28±7 days after the final dose of IMM-101.
- 5. During the Maintenance Phase of the study, in the event of an injection site reaction ≥Grade 3 (severe) as measured by the NCI CTCAE v4.0<sup>[⊥]</sup>, or at the discretion of the Investigator, patients may be administered a half dose of IMM-101 (0.5 mg/0.05 mL) or the dosing interval may be increased <u>or both</u>. If the dosing interval is increased, the patient should attend the study site for safety assessments at least every 14 weeks.
- 6. A full physical examination will be performed. Any additional physical examinations to those scheduled for this study will be performed as per the Investigator's routine procedures.
- 7. Any additional blood tests to those scheduled will be performed as per the Investigator's routine procedures.
- 8. Prior to administration of IMM-101.
- 9. Blood and serum samples (6 mL blood) CRP, FBC (Hb, haematocrit, RBC count, WBC count, WBC differential count, platelet count, MPV, MCV, MCH), LFTs (ALT, ALP, AST, bilirubin [total, direct], albumin, total protein, GGT, Pt/PTT, INR, LDH), calcium, urea and electrolytes (kidney function: sodium, potassium, creatinine, urea, eGFR [using CKD-EPI creatinine calculation]), CEA and CA19.9.
- 10. Patients in the anti-PD1 and anti-CTLA-4 cohorts only, prior to every course of checkpoint inhibitor as per the label: thyroid function test; ACTH; blood glucose test; lipase.
- 11. Every 14 weeks or as close to this time frame as possible.
- 12. Patients in the anti-PD1 and anti-CTLA-4 cohorts only: thyroid function test; ACTH; blood glucose test; lipase.
- 13. Immunological markers:
  - 6 mL whole blood: miRNA panel, circulating metabolites.
  - 6 mL whole blood will be collected from a subset of patients for FACS analysis: immune cell quantification.
  - 6 mL whole blood will be collected from a subset of patients to be analysed in the TruCulture system: cytokines, chemokines, immune mediators; functional immune cell assays, tumour markers.
- 14. Resting blood pressure, pulse, and body temperature will be recorded as vital signs at the EOS visit. Additional measures of vital signs to those scheduled for this study will be performed as per the Investigator's routine procedures.
- 15. Additional 12-lead ECG measures to those scheduled for this study will be performed as per the Investigator's routine procedures.
- 16. Two observers will be required to assess performance status. If there is any discrepancy between the two scores, the highest (worst) assessment will be used
- 17. Scans performed to assess progression or response must match the baseline scan (i.e. if CT scan at baseline then CT scan for all other scans). Additional CT/MRI scans to those scheduled for this study will be performed as per the Investigator's routine procedures.
- 18. Only required if no scan has been performed in the 6 weeks prior to the EOS visit.
- 19. All prescription and over-the-counter medications, including herbals, homeopathic remedies etc. will be recorded.
- 20. All AEs will be followed until resolution, death, or 30 days after the Withdrawal/EOS visit (whichever comes first)
- 21. Solicited and visible injection site reactions will be recorded.


#### 5.2 Study Data Sets

The definitions of the data sets for the IMM-101-011 study are given below.

#### 5.2.1 All Enrolled Patients

Enrolled patients are patients who enter the study at Visit 1 Day 0, following completion of screening assessments and confirmation of eligibility to enter the study. All listings are based on this set of patients. Hence data for the patient who failed screening will not be listed.

### 5.2.2 Safety Analysis Set (SAF)

The safety analysis set (SAF) includes all patients who took at least one administration of study treatment (IMM-101).

#### 5.3 Withdrawn Patients

Details of withdrawal procedures are described in the study Protocol.

On 31<sup>st</sup> July 2017, Immodulon took the decision to enroll no further patients into this Phase I/IIa open-label study and to close the study early. Hence, the 2 enrolled patients who were on study at this date both completed their withdrawal visit in place of Visit 6 – Week 12. Their last study visit completed was Visit 5 – Week 10 for both patients.

#### 5.4 Randomisation

Not applicable.

## 5.5 **Blinding**

Not applicable.

## 5.6 Sample Size

The study was terminated by the sponsor and the two enrolled patients were withdrawn. The last study visit completed was Visit 5 – Week 10. The End of Study / Withdrawal Visit was completed in place of Visit 6 – Week 12 for both patients.

## 5.7 Changes in Conduct or Planned Analyses from the Protocol

Due to the early termination of the study with only 2 enrolled patients, both of whom were withdrawn early, the objectives of the study could not be met. Hence the planned analyses described in the study Protocol will not be carried out. However, the data collected in the eCRF will be listed.

## 6 Statistical Methodology

## 6.1 Planned Presentations of Data: Listings

The presentation of listings and conventions for the listings are contained in a separate document. Both this SAP and the listings shells document will be approved before database lock.

This section therefore provides a tabular summary of the planned listings including listing number, title, medical coding dictionary data (and version), additional derived data and details of derivation.

All patient data will be presented in separate data listings by data type.

#### 6.1.1 Standard Calculations

Study day will be calculated as visit number date (or date of assessment/date of finding/AE/medication etc.) - date of Day 0 (first study drug administration dosing date) and will appear on all relevant dates throughout the listings. Day numbers prior to first study drug administration dosing date (for example screening assessments) will therefore be represented by a negative number of days.

The baseline value (for change from baseline calculations) will be defined as the last assessment prior to the first administration of study drug. The baseline value will be the Screening value if there is no Visit 1 day 0 value.

| Listing number | Listing title | Medical dictionary coding items | Derived data | Derivation |
|---|---|---|---|---|
| 16.2.1.1 | Patient Completions and Withdrawals | | Time on study (months) | (Date of study withdrawal – date of Day 0 +1 day)/30.4375 |
| 16.2.2.1 | Protocol Deviations | | | |
| 16.2.2.2 | Eligibility | | | |
| 16.2.2.3 | Informed Consent | | | |
| 16.2.3.1 | Analysis Sets | | SAF | All patients who took at least one administration of study treatment (IMM-101). |
| 16.2.4.1 | Demography | | Age (years) | Age is calculated in years from the date of informed consent, as the number of full months between date of birth and informed consent divided by 12 and rounded to the lowest integer. |
| | | | Body Mass<br>Index (kg/m²) | Weight (kg)/height (m)^2). |


| 16.2.4.2 | Medical History (Other Than Cancer History) | Medical history will be coded using the Medical Dictionary For Regulatory Activities (MedDRA) version 20 | | |
|---|---|---|---|---|
| 16.2.4.3 | Cancer Diagnosis | Cancer diagnoses<br>will be coded<br>using MedDRA<br>version 20 | Time since diagnosis (months) | (Day 0 (i.e. first study medication administration date) - date of diagnosis + 1)/30.4375 |
| 16.2.4.4 | HLA Serotyping at Screening | | | |
| 16.2.4.5 | Serum Pregnancy Test | | | |
| 16.2.4.6 | Microsatellite Phenotyping at Screening | | | |
| 16.2.4.7 | Prior and Concomitant Medications (Excluding Cancer Medications) | Medications will<br>be coded using<br>WHO Drug<br>Dictionary, version<br>September 2017 | | |
| 16.2.4.8 | Standard of Care Therapy | Medications will<br>be coded using<br>WHO Drug<br>Dictionary,<br>September 2017 | | |


| 16.2.4.9 | New Cancer Medications (Post-standard of Care) | Medications will<br>be coded using<br>WHO Drug<br>Dictionary, version<br>September 2017 | | |
|---|---|---|---|---|
| 16.2.4.10 | Radiotherapy | | | |
| 16.2.4.11 | Cancer-related Surgery | | | |
| 16.2.5.1 | Study Drug Administration | | Duration of exposure (days) | Date of last study<br>treatment administration –<br>date of first study<br>treatment administration +<br>1 |
| 16.2.6.1 | Tumour Biopsy - Core Samples | | | |
| 16.2.6.2 | Target Lesions | | | |
| 16.2.6.3 | Non-target Lesions | | | |
| 16.2.6.4 | Target Lesion Response to Treatment | | | |
| 16.2.6.5 | Overall Response to Treatment | | | |
| 16.2.7.1 | Adverse Events | Adverse events<br>will be coded<br>using MedDRA<br>version 20 | Treatment<br>emergent | An adverse event that started after administration of study drug |
| | | | Time to onset | Time from date of first administration of study |


| | | (d:hh:mm) | drug to onset of adverse event. Note: For missing or partial dates and times, not calculated and is reported as unknown (UK). |
|---|---|---|---|
| 16.2.8.1.1 | All Haematology Values | Change from baseline | Value at assessment time point – baseline value |
| | | H, L | Above normal range, below normal range |
| 16.2.8.1.2 | Patients with Clinically Significant Haematology Values | H, L | Above normal range, below normal range |
| 16.2.8.2.1 | All Biochemistry Values | Change from baseline | Value at assessment time point – baseline value |
| | | H, L | Above normal range, below normal range |
| 16.2.8.2.2 | Patients with Clinically Significant Biochemistry Values | H, L | Above normal range, below normal range |
| 16.2.9.1 | Immunology Sampling | | |
| 16.2.9.2 | Injection Site Reactions | | |
| 16.2.9.3 | Vital Signs | Change from baseline | Value at assessment time point – baseline value |
| 16.2.9.4 | Weight | Change from | Value at assessment time |


| | | baseline | point – baseline value |
|---|---|---|---|
| 16.2.9.5 | ECG Results | Change from baseline | Value at assessment time point – baseline value |
| 16.2.9.6 | Physical Examination | | |
| 16.2.9.7 | ECOG/WHO Performance Status | Highest (worst) Maximum ECOG/WHO performance status | Maximum score of the first and second evaluators' assessments |
| 16.2.9.8 | Diameter of Erythema and Skin Biopsy | | |


## 6.2 Adjustment for Covariates

Not applicable.

#### **6.2.1 Centre Effects**

Not applicable.

#### 6.3 **Protocol Violations**

Protocol deviations are recorded in the eCRF and presented in a data listing.

## 6.4 Missing Values – Missing Visits

There is no intention to implement any procedure for replacing missing data, other than as specified in this SAP.

## 6.5 Deviations from Statistical Analysis Plan

All deviations from this approved SAP will be described and justified in the final CSR. No pre-database lock data review meeting will be held, however the data will be reviewed by Immodulon prior to database lock.